CLINICAL TRIAL: NCT06887426
Title: Cladribine Tablets as an Exit Therapy Strategy: Alternative to Continuing Treatment and Plain Treatment Discontinuation in Ageing Stable RMS Patients
Brief Title: Cladribine Tablets as an Exit Therapy Strategy
Acronym: CLADREXIT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9628
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Cladribine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cladribine group
  Interventions: Drug: Cladribine
- Continuing treatment group

INTERVENTIONS:
Drug: Cladribine — To evaluate the clinical activity during the 2 years of follow-up in patients switching to cladribine and continuing current DMT
  Groups: Cladribine group

SUMMARY:
The objective of the study is to evaluate the effectiveness of CladT, in terms of disease stability and safety, as the last treatment option in ageing MS patients vs treatment continuation and discontinuation This observational study will use database from local cohorts (from France, Belgium, Switzerland). Patients included must meet the inclusion criteria: RRMS diagnosis for more than 10 years without secondary progression, no evidence of disease activity (no relapse, no new MRI lesion, no EDSS progression) for more than 5 years under a DMT, age≥ 45-year-old.

Analyses will be using dynamic propensity score to match patients who stopped treatment with patients who had the same probability of continuing / stopping current treatments but took CladT as exit therapy. Patients with a minimum of 24 months follow up will be included.

The investigators will ensure that CladT provide disease stability compared to treatment continuation / discontinuation in ageing MS patients by measuring:

* the percentage of patients free of relapse, and time to first relapse, defined as the appearance, recurrence, or aggravation of neurological symptoms for a period of at least 24 hours without fever.
* the percentage of patients free of EDSS progression confirmed for at least 6 months and until the end of patient follow up.
* the percentage of patients free of MRI activity, defined as new or enlarged T2 lesions compared with the previous brain MRI scan or gadolinium enhancing T1 lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥45-year-old with RRMS
* Disease duration ≥10 years
* No evidence of disease activity ≥5 years under DMT
* EDSS score between 0 and 6.0 included

Exclusion Criteria:

* Progressive form of MS
* Patients without DMT
* EDSS score ≥6.5

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicentric retrospective and controlled cohort with non-inferiority analysis. Patients will be matched 1:1 using propensity score on gender, age, MS duration, time before last relapse, EDSS score, DMTs.
  The study will use retrospectively collected data within the date frame from 06/30/25 to 06/30/26.
  Approximately 150 patients treated with cladribine will be identified and included in this study in 7 centers: Strasbourg, Lille, Montpellier, Nimes, Liège, Pelt, Lugano.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical activity during the 2 years of follow-up in patients switching to cladribine and continuing current DMT | 2 years
  Proportion of patients with relapses* and time to event during the 2 years of follow-up in patients switching to cladribine and continuing current DMT

SECONDARY OUTCOMES:
To evaluate the clinical activity during the 2 years of follow-up in patients switching to cladribine and stopping current DMT | 2 years
  Proportion of patients with relapse and time to event during the 2 years of follow-up in patients switching to cladribine and stopping current DMT
To evaluate the clinical activity during the 3 years of follow-up in patients switching to cladribine and continuing current DMT | 2 years
  Proportion of patients with relapse and time to event during the 2 years of follow-up in patients switching to cladribine and continuing current DMT
To evaluate the radiological activity during the follow-up in patients switching to cladribine, continuing current DMT and stopping DMT | 2 years
  Proportion of patients with new T2 lesions on brain MRI at 1 and 2 years in patients switching to cladribine, continuing current DMT and stopping DMT
To evaluate the disability during the follow-up in patients switching to cladribine, continuing current DMT and stopping DMT | 2 years
  Proportion of patients with EDSS worsening** after 2 years in patients switching to cladribine, continuing current DMT and stopping DMT
To evaluate the risk of serious adverse events in patients switching to cladribine and continuing current DMT | 2 years
  Proportion of patients with any serious adverse events after 2 years in patients switching to cladribine and continuing current DMT

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie - Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided